CLINICAL TRIAL: NCT02587637
Title: A Prospective Post Market Observational Pilot Study to Evaluate the Effectiveness of DRG Stimulation in the Treatment of Discogenic Low Back Pain
Brief Title: Study to Evaluate the Effectiveness of DRG Stimulation for Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28-SMI-2015
Record Dates: First submitted 2015-10-22; First posted 2015-10-27 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Chronic Pain
Keywords: Chronic Low Back Pain; Dorsal Root Ganglion; Neurostimulator System; spinal cord stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single device arm (Other)
  Interventions: Device: Dorsal root ganglion (DRG) stimulation

INTERVENTIONS:
Device: Dorsal root ganglion (DRG) stimulation — The role the DRG plays in the development and maintenance of chronic pain, we have developed a neurostimulator system for the management of chronic intractable pain by electrically stimulating the DRG

SUMMARY:
The purpose of this prospective post market observational pilot study is to evaluate the effect of DRG stimulation in the management of chronic discogenic pain in subjects who are refractory to other available treatments. Selected subjects will not be suitable candidates for lumbar spinal surgery and will meet the standard selection process for DRG stimulation as routinely utilised in the study centre. Results from this pilot study will inform current clinical practice and future comparative studies in this specific population.

ELIGIBILITY:
Inclusion Criteria:

1. Subject of either gender between 18 and 65 years of age
2. Subject is able and willing to comply with the follow-up schedule and protocol
3. Subject is able to provide written informed consent
4. Chronic low back pain of at least 6 months
5. History consistent with discogenic low back pain (e.g. Pain produced on lumbar motion, significant functional limitation in sitting duration and tolerance)
6. Neurologic exam without marked motor deficit.
7. Definite/Highly Probable/Discogenic Pain as confirmed by provocative discography according to IASP/ISIS guidelines*
8. Low Back Pain intensity should be 6 or higher measured on a NPRS at baseline
9. Meets all the inclusion criteria for the implantation of a neurostimulation system as typically utilised in the study centre
10. Subject has been screened by a multi-disciplinary panel including a psychologist and deemed suitable for implantation

Exclusion Criteria:

1. Female subject of childbearing potential is pregnant/nursing or plans to become pregnant during the course of the study
2. Escalating or changing pain condition within the past month as evidenced by investigator examination
3. BMI ≥35
4. Subject has had injection therapy or radiofrequency treatment for their low back pain within the past 3 months
5. Subject currently has an active implantable device including ICD, pacemaker, spinal cord stimulator or intrathecal drug pump
6. Subject is unable to operate the device
7. Severe disc degeneration at the affected level as evidenced by >50% disc height loss on plain anteroposterior and lateral lumbar radiographs or CT/MRI.
8. Extruded or sequestered herniated nucleus pulposus at the affected level(s).
9. Previous lumbar back surgery (e.g. Laminectomy, discectomy or fusion) at the affected level(s)
10. Moderate to severe spinal stenosis due to osteophyte and/or ligamentous overgrowth as evidenced by MRI or CT in the previous 6 months
11. Moderate to severe endplate degenerative changes at the affected levels
12. Grade 1-2 spondylolisthesis
13. Previous Neurostimulation therapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Ziekenhuis, Velp, Velp, Arnhem, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- All Subjects: Subjects with confirmed discogenic low back pain enrolled in the study
Period: Overall Study
Arm/Group | All Subjects
Started | 20
Received Intervention | 15
Completed | 14
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Subjects
Number analyzed (Participants) | 20
Age, Customized [Mean (Full Range); unit: years] — between 22 and 71 years of age
  years | 45 [22 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Netherlands | 20

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With 30% or Greater Reduction in Back Pain at 6 Months
Description: The number (percentage) of subjects who achieve a sustained and clinically meaningful reduction in the intensity of LBP of ≥30% or 2 points on a numerical pain rating scale (NPRS) in the implanted subjects at 6 month follow-up visit as compared to baseline.
Time Frame: 6 months
Population: 15 patients were implanted with the DRG Axium system.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants | 11

2. Primary Outcome: Percentage of Subjects With 30% or Greater Reduction in Back Pain at 12 Months
Description: The number (percentage) of subjects who achieve a sustained and clinically meaningful reduction in the intensity of LBP of ≥30% or 2 points on a numerical pain rating scale (NPRS) in the implanted subjects at 12 month follow-up visit as compared to baseline.
Time Frame: 12 months
Population: 15 patients were implanted with the DRG Axium system, 14 patients have available data for pain relief at 12 months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Participants | 13

3. Secondary Outcome: Percentage of Patients With Improved Global Impression of Change at 6 Months
Description: The subject was requested to rate their overall change in activity limitations, symptoms, emotions and overall quality of life related to his/her condition on a seven-point categorical scale (much worse, worse, somewhat worse, no change, slightly better, better and much better). Patients who reported to be much better or better are counted.
Time Frame: 6 Months
Population: 15 patients had available data at 6 Months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants | 10

4. Secondary Outcome: Percentage of Patients With Improved Global Impression of Change at 12 Months Using Trial System
Description: as for outcome 3
Time Frame: 12 Months
Population: 14 patients had available data at 12 Months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Participants | 11

5. Secondary Outcome: Percentage of Subjects With 50% or Greater Reduction in Back Pain at 6 Months
Description: Subjects experiencing 50% or more reduction in the intensity of the back pain.
Time Frame: 6 Months
Population: 15 patients had available data at 6 Months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 15
Participants | 11

6. Secondary Outcome: Percentage of Subjects With 50% or Greater Reduction in Back Pain at 12 Months
Description: Subjects experiencing 50% or more reduction in the intensity of the back pain.
Time Frame: 12 Months
Population: 14 patients had available data at 12 Months.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 14
Participants | 11

ADVERSE EVENTS:
Time Frame: device related AE's and SAE's were reported from Informed Consent signature until the last follow-up visit (12 Months)
Description: Only device related AE's and SAE's were reported
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=20)
Increased Pain (General disorders) | 5 (5)
Pain at pocket (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-19): https://cdn.clinicaltrials.gov/large-docs/37/NCT02587637/Prot_SAP_000.pdf